CLINICAL TRIAL: NCT00403208
Title: Clinical and Economical Impact of an Analgesia-Based, Goal-Directed, Nurse-Driven Sedation Protocol on Patients on Mechanical Ventilation. A Multicenter Study
Brief Title: Analgesia-Based Sedation During Mechanical Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SA05I20091
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Last update posted 2006-11-28 (Estimated); Status verified 2006-11

CONDITIONS: Ventilation, Mechanical; Respiratory Insufficiency; Critical Illness
Keywords: Ventilation, Mechanical; Sedation
MeSH Terms: conditions — Respiratory Aspiration; Respiratory Insufficiency; Critical Illness

INTERVENTIONS:
Procedure: Analgesia based sedation in ICU patients

SUMMARY:
Hypothesis: A protocolized algorithm for sedation in critically ill patients on mechanical ventilation can decrease ventilator days, costs and improve outcome.

This is a multicenter observational-interventional study on critically ill patients who require mechanical ventilation for more than 48 hours, involving 13 ICU in Chile. There are two periods (groups): a descriptive phase of sedation practices, and an interventional period in which an analgesia-based, goal-directed, nurse-driven sedation is applied.

Main outcome: ventilator-free days between both periods.

DETAILED DESCRIPTION:
This is a multicenter observational-interventional study on critically ill patients who require mechanical ventilation for more than 48 hours, involving 13 ICU in Chile.

Main exclusion criteria are neurologic impairment, previous chronic cardiac, liver and renal failure, second period of mechanical ventilation during hospitalization, short term expected mortality.

There is an initial descriptive phase of sedation practice, involving sedative drugs, sedation level assessment, and outcome: ventilator-free days, ICU stay, costs and mortality.

After a period of analysis and training, an analgesia-based, goal-directed, nurse-driven sedation protocol is applied. Fentanyl infusion is started and titrated to obtain a patient calm and cooperative or mildly sedated while on mechanical ventilation. Hypnotics and opiates i.v. boluses are allowed during the first hours of mechanical ventilation. Midazolam infusion is started if ventilatory distress continue despite fentanyl 1.8 µg/kg/min. Haldol, muscle relaxants and other sedative drugs are allowed depending on patient condition. After 48 hours of mechanical ventilation, sedative drugs are discontinued in the morning.

Main outcome: ventilator-free days. Secondary outcome: ICU stay, costs, and sedation quality. At 6 moths SF-36. Each period is planned to included at least 140 patients, for a 20% difference in ventilator-free days, with 80% power and a 0.05 type I error.

ELIGIBILITY:
Inclusion Criteria:

* Patients who require mechanical ventilation for more than 48 hours

Exclusion Criteria:

* Nervous system diseases
* Previous liver or renal failure
* Second episode of MV during same hospitalization
* Expected MV shorter than 48 hours
* Short term expected mortality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280
Dates: Start 2006-03; Study Completion 2006-11

PRIMARY OUTCOMES:
Ventilator-free days

SECONDARY OUTCOMES:
ICU stay
ICU cost
Sedation quality
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Bugedo, MD, Principal Investigator — Universidad Catolica de Chile
Locations (14):
- Chile (14):
  - Hospital Regional de Coquimbo, Coquimbo
  - Hospital Universidad Catolica de Chile, Santiago
  - Clinica Alemana, Santiago
  - Hospital Clinico Universidad de Chile, Santiago
  - Hospital Dipreca, Santiago
  - Hospital Luis Tisne, Santiago
  - Hospital Militar, Santiago
  - Hospital Padre Hurtado, Santiago
  - Hospital San Jose, Santiago
  - Hospital San Juan de Dios, Santiago
  - Hospital Sotero del Rio, Santiago
  - Hospital Regional de Talca, Talca
  - Hospital Carlos Van Buren, Valparaíso
  - Hospital Naval, Viña del Mar